CLINICAL TRIAL: NCT02244242
Title: A Forty-Five Day, Open-label Study of the Symptomatic Relief Effects of FLOMAX® Capsules 0.4 mg Daily in Patients With the Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Study to Evaluate the Symptomatic Relief Effects of FLOMAX® in Patients With Signs and Symptoms of Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 527.16
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

ARMS (1):
- Tamsulosin hydrochloride (Experimental): modified release capsules
  Interventions: Drug: Tamsulosin hydrochloride

INTERVENTIONS:
Drug: Tamsulosin hydrochloride
  Other Names: Flomax®

SUMMARY:
Study to evaluate the symptomatic relief afforded by tamsulosin hydrochloride capsules in patients with signs and symptoms of benign prostatic hyperplasia (BPH). Additionally to provide primary care physicians experience with the use of tamsulosin hydrochloride capsules 0.4 mg daily for the treatment of BPH

ELIGIBILITY:
Inclusion Criteria:

* Male patients (45 years of age or older) diagnosed with BPH who scores at least 13 points on the AUA Symptom Score Index at baseline
* Patients who have a baseline Prostate specific antigen (PSA) of >= 4.0 ng/ml
* Patients who provide written informed consent prior to participation in the study in accordance with regulatory requirements
* Patients who have been judged by the investigator to be reliable and who have agreed to cooperate with all tests and examinations stipulated in the protocol

Exclusion Criteria:

* Patients who have previously been diagnosed with prostate cancer
* Patients who have an abnormal Digital rectal examination (DRE) of the prostate gland at baseline other than enlargement (i.e., patients with suspicious areas or nodularity of the gland which may indicate possible prostatic carcinoma are to be excluded)
* Patients who have had previous invasive or non-invasive surgical treatment of the prostate gland
* Patients who have had an episode of acute urinary retention within four weeks of the screening visit
* Patients who have a history or evidence of urethral stricture
* Patients who have had pelvic radiotherapy
* Patients who have a history of chronic prostatitis
* Patients who have a history of neurogenic bladder
* Patients who have had a urinary tract infection (i.e. positive urine culture yielding pathogenic bacteria >= 10**5 colony forming units per ml or a laboratory report of a urinary tract infection) or symptoms/signs indicative of a urinary tract infection such as: increased white blood cells (WBCs) in the urine (15-30 WBC/high powered field [hpf], dysuria, costovertebral tenderness and urinary frequency accompanied by fever within four weeks of baseline
* Patients who have evidence of significant renal dysfunction based upon a serum creatinine greater than two times the upper limit of normal levels established by the central laboratory used in this study
* Patients who have baseline clinical laboratory test results that indicate the following values:

  * Hemoglobin: < 12.0 g/dl
  * Leukocytes: < 3000 mm³
  * Liver enzymes: Serum Glutamic Oxaloacetic Transaminase (SGOT), Serum Glutamic Pyruvic Transaminase (SGPT), Gamma-Glutamyl Transferase (GGT) and alkaline phosphatase): More than two times the upper limit of normal levels established by the central laboratory used in the study
* Patients who have postural symptoms (e.g. lightheadedness, dizziness and fainting occurring with or without a change in Blood Pressure (BP) and/or Heart Rate (HR) within four weeks of baseline
* Patients who have participated in another drug study within four weeks of baseline
* Patients who have clinically relevant conditions which might interfere with the patient's ability to participate in the study including (but not limited to) the following:

  * neurologic, gastrointestinal, cardiovascular (including uncontrolled hypertension defined as a sitting diastolic BP >= 95 mmHg with or without treatment), hepatic, renal, psychiatric, hematologic or respiratory disease or clinically relevant laboratory abnormalities based upon the investigator's judgment
* Patients who have had cancer or a diagnosis of cancer within five years of baseline
* Patients who have received cimetidine, warfarin or herbal medication specifically for treatment of any urological problems within four weeks prior or baseline
* Patients who have known allergy to study medication
* Patients who are currently receiving finasteride or who have been treated with finasteride within three months prior to baseline
* Patients who have documented myocardial infarction (by ECG) within the past 6 months or evidence of a myocardial infarction on an ECG where the date could not be determined
* Patients who are classified as New York Heart Association (NYHA) Class III or IV congestive heart failure
* Patients who have prosthetic heart valves, cardiac devices or history of endocarditis
* Patient who have clinically significant cardiac arrhythmias as diagnosed by ECG whether or not accompanied by symptoms (e.g., dizziness, presyncope, syncope, unsteadiness)
* Patients who have received the following drugs within two weeks prior to baseline and who are unable to discontinue these drugs for the remainder of the study:

  1. Alpha-adrenergic blocking agents
  2. Alpha-adrenergic agonists
  3. Drugs with anticholinergic activity including antihistamines
  4. Antispasmodics
  5. Parasympathomimetics and cholinomimetics

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 1998-07; Primary Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Change in American Urological Association (AUA) Symptom Score Index by means of a patient self-assessment questionnaire | up to 45 days

SECONDARY OUTCOMES:
Change of AUA Bother Score Index by means of a patient self-assessment questionnaire | up to 45 days
Change in BPH Impact Index by means of a patient self-assessment questionnaire | up to 45 days
Global Assessment of investigator on 5-point scale | at 4, 8 and 45 days
Number of patients with adverse events | up to 59 days